CLINICAL TRIAL: NCT05170243
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics Characteristics and Immunogenicity of a Single Dose of 9MW1911 Injection in Healthy Subjects
Brief Title: A Clinical Study in Healthy Subjects to Evaluate 9MW1911 Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9MW1911-2021-CP102
Record Dates: First submitted 2021-12-12; First posted 2021-12-27 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Asthma; COPD; Atopic Dermatitis
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 9MW1911 Injection (Active Comparator): Experimental drug administered IV infusion
  Interventions: Drug: 9MW1911 Injection
- 9MW1911 Injection Placebo (Placebo Comparator): Placebo administered IV infusion
  Interventions: Drug: 9MW1911 Injection Placebo

INTERVENTIONS:
Drug: 9MW1911 Injection — Single dose intravenously on day 1
  Arms: 9MW1911 Injection
Drug: 9MW1911 Injection Placebo — Single dose of matching placebo intravenously on day 1
  Arms: 9MW1911 Injection Placebo

SUMMARY:
This is a Phase 1, randomized, placebo-controlled study, enrolling approximately 38 healthy adult subjects (18-65 yrs). The purpose of this study is to evaluate the safety, tolerability and PK of single ascending dose of 9MW1911 administered intravenously (IV) in healthy adult volunteers. All subjects will be followed up for safety from the time of Informed Consent through 113 days post dose.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are willing to follow study procedures and sign informed consent voluntarily.
2. Male or female subjects aged 18 to 65 years (including 18 and 65 years).
3. Weight≥50.0 kg for males, or weight≥45.0 kg for females, and body mass index (BMI) in the range of 19.0 ~ 26.0 kg/m2 (including cut-off value).
4. Female subjects must have a negative β-HCG pregnancy test (Screening and Baseline); Subjects(including their partners) will take effective contraceptive measures voluntarily;Subjects have neither pregnancy plans nor sperm or egg donation plans during the screening period and the next 6 months.

Exclusion Criteria:

1. Subjects who have a history of allergies to biological agents or any drug components; those who have a history of allergies and judged by the investigator to be ineligible for enrollment.
2. The clinical laboratory tests show any clinical abnormalities, or abnormalities with clinical significance(including but not limited to diseases of digestive tract, kidney, liver, nervous system, blood, endocrine system, cancer, lung, immune system, mental, heart),and judged by the investigator to affect participation in this study.
3. Subjects with prolonged QTcF interval (> 450 ms) on electrocardiogram (ECG) examination, or family history of prolonged QTc syndrome or sudden death.
4. Subjects (female) who is pregnant or lactating at screening or during the trial.
5. Subjects who have previously used immunosuppressants or monoclonal antibodies for any reason.
6. Subjects who used any prescription, over-the-counter, or Chinese herbal medicines within 2 weeks prior to screening.
7. Subjects who received any vaccinations within 4 weeks prior to screening, or are scheduled to receive a vaccination during the study.
8. Subjects who have undergone surgery within 3 months prior to screening, or plan to undergo surgery during the study.
9. Subjects who have a history of drug abuse within 6 months prior to screening.
10. Subjects who have used illicit drugs within 3 months prior to screening.
11. Subjects who have consumed more than 14 units of alcohol per week (1 unit of alcohol ≈ 360 mL of beer or 45 mL of spirits containing 40% alcohol or 150 mL of wine) within 3 months prior to screening, or who cannot abstain from alcohol during the study.
12. Subjects who have smoked more than 5 cigarettes per day within 3 months prior to screening, or who cannot abstain from cigarette product during the study.
13. Subjects who have participated in drug or medical devices clinical trials within 3 months prior to screening.
14. Subjects who donated or lost blood ≥ 200 mL within 3 months prior to screening, or plan to donate blood within 3 months.
15. Subjects whose alcohol breath test results greater than 0.0 mg/100 ml or positive drug screening (morphine, icenarcotics [methamphetamine], ketamine, ecstasy [methylenedioxyamphetamine], cannabis [tetrahydrocannabinolate]).
16. Subjects who have one or more clinically significant tests of hepatitis B virological markers, hepatitis C virus antibodies, anti-human immunodeficiency virus antibodies, or anti-Treponema pallidum-specific antibodies.
17. Subjects who cannot tolerate venipuncture or have a history of needle-sickness and blood-sickness.
18. Subjects who show insufficient communication, understanding and cooperation, or poor compliance to ensure observation and follow-up as required by the protocol.
19. Subjects with abnormal vital signs with clinical significance: diastolic blood pressure≤50 mmHg or ≥90 mmHg, pulse≤50 beats/min or ≥100 beats/min, body temperature (ear temperature) <35.5°C or >37.5°C, respiration>20 breaths/min. The specific situation will be comprehensively determined by the investigator.
20. Subjects who is inappropriate to participate in the trial due to any reasons as determined by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-07-03 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Adverse Event(including serious adverse event) | up to day 113
  The incidence of AEs (adverse events) and SAEs (serious adverse events) from treatment until the last scheduled follow-up visit

SECONDARY OUTCOMES:
PK parameters | up to day 113
  Maximum concentration(Cmax)
PK parameters | up to day 113
  The area under the curve (AUC)
PK parameters | up to day 113
  Time at which maximum concentration(Tmax)
PK parameters | up to day 113
  The half life(T1/2)
Incidence of ADAs Against 9MW1911 | up to day 113
  The incidence of ADAs against 9MW1911 during the study will be summarized

CONTACTS AND LOCATIONS:
Overall Officials: Wang Shuhai, Ph.D, Study Chair — Mabwell (Shanghai) Bioscience Co., Ltd.
Locations (1):
- Shanghai Public Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No